# Informed consent

Social Media and Suicidal Behavior: A Study on the Impact of Journalistic Posts about Suicide on Commentators and Readers – Study 1 Dear Sir/Madam,

Thank you for your willingness to participate in the research. Please take a moment to read some important information about the study and its procedures.

About the project "Social Media and Suicidal Behavior: A Study on the Impact of Journalistic Posts about Suicide on Commentators and Readers" and the specific research:

Numerous studies indicate that inappropriate journalistic reporting on suicide can increase the risk of imitating reported behavior, while responsible reporting protects against imitation and encourages the search for more constructive ways to cope. However, there is limited research exploring the connection between online journalistic reporting on suicide and suicidal behavior in the population. There are even fewer studies on the role and characteristics of posts on suicide by journalists on social media and comments under these posts, as well as the correlation of these with the user's experience of these posts. This gap is addressed in this project.

#### **Research Purpose:**

The aim of this study is to examine the characteristics of journalistic posts on suicide published on social networks. Based on identified features, we aim to explore the impact of these posts on the user's experience and develop guidelines for responsible reporting and commenting on the topic of suicide on social media.

#### **Study Procedure:**

The entire project runs from October 1, 2021, to September 30, 2024. In the first part of the study, we began by examining the characteristics of journalistic posts on suicide published on social networks and comments under these posts. In the second part of the study, to which we also invite you, completing online questionnaires will follow, focusing on your psychological well-being, possible symptoms of depression, and the presence of suicidal thoughts. If you meet the inclusion criteria for participation in the study, you will be invited to review various posts on suicide by journalists on social networks (on the topic of suicide, traffic accidents, or posts related to weather phenomena). The review of posts will take place live, with a small number of other participants and a researcher from the UP IAM Slovenian Center for Suicide Research present. Your task will be to view the posts and answer questions related to your experience and mood. The estimated duration of the first measurement is approximately 10-15 minutes, and the second is 35 minutes. We have obtained ethical consent from the UP Ethics Committee for research involving human subjects.

## **Benefits of Your Participation:**

Your responses in the study will help us understand how journalistic reporting on suicide on social media affects the experience of other social media users. Based on this, we will formulate guidelines for reporting on suicide on social media. Additionally, participants in the second measurement will receive compensation in the form of a voucher worth 10 euros for a grocery store.

## **Voluntary Participation and the Option to Withdraw:**

Participation in the study is entirely voluntary, and you can withdraw at any time without any consequences.

## Risks to You and Your Health in Participation:

The study will present more and less appropriate posts on the topic of suicide, traffic accidents, and posts related to weather phenomena, and we will be interested in your personal experience. As some discomfort may arise, we will provide a debriefing conversation to all research participants after the measurement and take action according to your needs. Participation in the study can be terminated at any time without additional explanations.

In case of discomfort or the desire to withdraw from participation, you can contact the researcher from UP IAM Slovenian Center for Suicide Research present at the measurement or at the email address info.scsr@upr.si or the support contacts listed on the link http://zivziv.si/sos/.

### What will happen to your data?

Due to data related to your mental health, we will collect personal information through which, in the case of very poor mental health or suicidal risk, we can recognize your identity and contact you to seek professional help. We will also contact you with further information based on this personal information when you meet the inclusion criteria for the experimental part of the study. Your personal data will be stored separately from the data collected in the study. Also, all collected data will be treated confidentially, meaning only researchers from UP IAM SCSR will have access to the data. The collected data will be stored in a secure electronic database of UP IAM SCSR for at least 10 years after the publication of the project results. All data will be used exclusively for educational and scientific research purposes and processed only at the group level. In case of your withdrawal from participation, all your data will be destroyed. After the publication of the research results, erasing data obtained during the research is no longer possible.

#### Where can you get more information about the research?

For additional information about the research and research findings, you can write to: <a href="mailto:info.scsr@upr.si">info.scsr@upr.si</a>.

Please indicate your agreement with the following:

- I have read the information about the research.
- I have read the information about the research.
- I am familiar with the purpose and procedure of the research.
- I am aware of the benefits and risks of this research.
- I am aware of the sources of assistance I can turn to in case of discomfort or distress.
- I had the opportunity to ask additional questions regarding the research.
- I understand which data will be collected and what will happen to my data.
- I understand that the data will be treated confidentially, and only researchers from UP IAM SCSR will have access to it.
- I allow my data to be used for educational and scientific research purposes.
- I am aware of the options for deleting my data.
- I understand that my participation in the research is voluntary, and I can withdraw at any time without consequences.

- I am aware of the possibility and method of communication with the researchers from UP IAM SCSR in case of additional questions and research findings.
- I allow researchers from UP IAM SCSR to contact me in case of additional questions related exclusively to this research.
- I understand the information provided in the invitation and agree to participate in the research.

Please enter your personal information in the boxes below, through which we can contact you regarding further steps in the research.

| Your full name: | |
|---|---|
| Your date of birth: | |
| Your email address: | |
| , , , | als of your name, the initials of your last name, day of<br>For example, Mojca Novak, born on September 5,<br>05NM): |

Thank you for your willingness to participate.

Principal Investigator: Prof. Dr. Diego de Leo

UP IAM Slovenian Center for Suicide Research

